CLINICAL TRIAL: NCT00885118
Title: A Phase II, Randomised, Double-blind, Placebo-controlled, Multiple Dose Study to Evaluate Pharmacodynamics, Pharmacokinetics, Safety, and Tolerability of Once Daily Oral Administration of BI 10773 (1 mg, 5 mg, 10 mg, and 25 mg) for 28 Days in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: 4 Weeks Treatment With Empagliflozin (BI 10773) in Japanese Type 2 Diabetic Patients (T2DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.15
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (5):
- BI 10773 low dose quaque die (QD) (Experimental): patient to receive a BI 10773 low dose tablet and a placebo tablet once daily
  Interventions: Drug: BI 10773; Drug: Placebo (low dose)
- BI 10773 mid-low dose QD (Experimental): patient to receive a BI 10773 middle dose tablet and a placebo tablet once daily
  Interventions: Drug: Placebo (middle dose); Drug: BI 10773
- BI 10773 mid-high dose QD (Experimental): patient to receive two tablets of BI 10773 middle dose once daily
  Interventions: Drug: BI 10773
- BI 10773 high dose QD (Experimental): patient to receive a BI 10773 high dose tablet and a placebo tablet once daily
  Interventions: Drug: BI 10773; Drug: Placebo (high dose)
- Placebo (Placebo Comparator): patient to receive two tablets of placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo (middle dose) — Placebo tablets once a day
  Arms: BI 10773 mid-low dose QD
Drug: Placebo — Placebo tablets once a day
  Arms: Placebo
Drug: BI 10773 — BI 10773 middle dose tablets once a day
  Arms: BI 10773 mid-high dose QD
Drug: BI 10773 — BI 10773 high dose tablets once a day
  Arms: BI 10773 high dose QD
Drug: BI 10773 — BI 10773 middle dose tablets once a day
  Arms: BI 10773 mid-low dose QD
Drug: Placebo (high dose) — Placebo tablets once a day
  Arms: BI 10773 high dose QD
Drug: BI 10773 — BI 10773 low dose tablets once a day
  Arms: BI 10773 low dose quaque die (QD)
Drug: Placebo (low dose) — Placebo tablets once a day
  Arms: BI 10773 low dose quaque die (QD)

SUMMARY:
The objective of this trial is to evaluate the pharmacodynamics, pharmacokinetics, safety, and tolerability of once daily oral administration of BI 10773 administered for 28 days in Japanese patients with T2DM.

ELIGIBILITY:
Inclusion criteria:

1. Japanese male or female patients with T2DM treated with diet and exercise alone or with one hypoglycaemic drug other than glitazones.
2. Hemoglobin A1c (HbA1c) at screening (Visit 1)

   * For patients treated with 1 other oral antidiabetic drug: HbA1c between 6.5% and 9.0%.
   * For patients not treated with any antidiabetic drug: HbA1c between 7.0% and 10.0%.
3. Age between 20 and 70 years
4. Body mass index (BMI) between18.0 and 40.0 kg/m2
5. Signed and dated written informed consent before admission to the trial in accordance with the Good Clinical Practice (GCP) and the local legislation.

Exclusion criteria:

1. Antidiabetic treatment with insulin or glitazones within 3 months before obtaining informed consent or with more than 1 oral hypoglycaemic agent at the time of informed consent
2. Fasted blood glucose of >240 mg/dL (>13.3 mmol/L) or a randomly determined blood glucose level of >400 mg/dL (22.2 mmol/L) on 2 consecutive days during wash-out period.
3. Myocardial infarction, stroke, or transient ischaemic attack within 6 months before informed consent.
4. Clinically relevant concomitant diseases other than T2DM, hyperlipidaemia, and medically treated hypertension before the first administration such as

   * Renal insufficiency (calculated estimated glomerular filtration rate <60)
   * Cardiac insufficiency of New York Heart Association (NYHA) II-IV or other known cardiovascular diseases including hypertension of >160/95 mmHg,
   * Neurological disorders (such as epilepsy) or psychiatric disorders
   * Acute or clinically relevant chronic infections (e.g., human immunodeficiency virus, hepatitis, repeated urogenital infections)
   * Any gastrointestinal, hepatic, respiratory, endocrine, or immunological disorder
5. Patients under treatment with any concomitant medication except for the following drugs at the time of informed consent.:

   * Statins.
   * Antihypertensives (diuretics not allowed)
   * alpha-Blockers for benign prostate hypertrophy
   * Occasional use of acetylsalicylic acid, ibuprofen, or paracetamol
6. Additional inclusion/exclusion criteria apply

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- Japan (5):
  - 1245.15.003 Boehringer Ingelheim Investigational Site, Hachioji, Tokyo
  - 1245.15.002 Boehringer Ingelheim Investigational Site, Koganei, Tokyo
  - 1245.15.001 Boehringer Ingelheim Investigational Site, Nakano-ku, Tokyo
  - 1245.15.005 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1245.15.004 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa

REFERENCES:
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Yasui A, Lee G, Hirase T, Kaneko T, Kaspers S, von Eynatten M, Okamura T. Empagliflozin Induces Transient Diuresis Without Changing Long-Term Overall Fluid Balance in Japanese Patients With Type 2 Diabetes. Diabetes Ther. 2018 Apr;9(2):863-871. doi: 10.1007/s13300-018-0385-5. Epub 2018 Feb 27. PMID 29488164
- [Derived] Kanada S, Koiwai K, Taniguchi A, Sarashina A, Seman L, Woerle HJ. Pharmacokinetics, pharmacodynamics, safety and tolerability of 4 weeks' treatment with empagliflozin in Japanese patients with type 2 diabetes mellitus. J Diabetes Investig. 2013 Nov 27;4(6):613-7. doi: 10.1111/jdi.12110. Epub 2013 Jun 25. PMID 24843716
- [Derived] Riggs MM, Staab A, Seman L, MacGregor TR, Bergsma TT, Gastonguay MR, Macha S. Population pharmacokinetics of empagliflozin, a sodium glucose cotransporter 2 inhibitor, in patients with type 2 diabetes. J Clin Pharmacol. 2013 Oct;53(10):1028-38. doi: 10.1002/jcph.147. Epub 2013 Aug 13. PMID 23940010

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Treatment with placebo once daily
- Empa 1 mg: Treatment with Empa 1 mg once daily
- Empa 5 mg: Treatment with Empa 5 mg once daily
- Empa 10 mg: Treatment with Empa 10 mg once daily
- Empa 25 mg: Treatment with Empa 25 mg once daily
Period: Overall Study
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Started | 21 | 19 | 21 | 20 | 19
Completed | 20 | 19 | 20 | 20 | 18
Not Completed | 1 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Other reason not defined above | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg | Total
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 19 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.0) | 58.6 (8.2) | 53.9 (9.9) | 55.8 (8.0) | 60.8 (8.7) | 57.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 1 | 3 | 4 | 16
  Male | 16 | 16 | 20 | 17 | 15 | 84

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Urine Glucose Excretion
Description: Change from baseline in Urine glucose excretion to 28 days
Time Frame: baseline and 28 days
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 20 | 19 | 20 | 18 | 17
mg | 599.763 (4497.460) | 43428.245 (4598.593) | 81564.440 (4460.086) | 89189.527 (4704.967) | 86220.111 (4828.541)
Statistical Analysis 1: Comparison: Placebo vs Empa 1 mg; Difference calculated as empa 1mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = 42828.482, 95% CI 2-sided [29936.586 to 55720.378], Standard Error of Mean 6487.174
Statistical Analysis 2: Comparison: Placebo vs Empa 5 mg; Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = 80964.677, 95% CI 2-sided [68437.160 to 93492.194], Standard Error of Mean 6303.820
Statistical Analysis 3: Comparison: Placebo vs Empa 10 mg; Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = 88589.764, 95% CI 2-sided [75583.738 to 101595.790], Standard Error of Mean 6544.604
Statistical Analysis 4: Comparison: Placebo vs Empa 25 mg; Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = 85620.348, 95% CI 2-sided [72484.181 to 98756.515], Standard Error of Mean 6610.091

2. Primary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Change from baseline in Fasting plasma glucose to 28 days
Time Frame: baseline and 28 days
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 20 | 19 | 20 | 18 | 17
mg/dL | -15.436 (2.860) | -28.116 (2.965) | -35.355 (2.865) | -41.643 (3.009) | -42.670 (3.089)
Statistical Analysis 1: Comparison: Placebo vs Empa 1 mg; Difference calculated as empa 1mg minus placebo; Test type: Superiority or Other; p = 0.0030, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -12.680, 95% CI 2-sided [-20.936 to -4.424], Standard Error of Mean 4.155
Statistical Analysis 2: Comparison: Placebo vs Empa 5 mg; Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -19.920, 95% CI 2-sided [-27.919 to -11.921], Standard Error of Mean 4.025
Statistical Analysis 3: Comparison: Placebo vs Empa 10 mg; Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -26.208, 95% CI 2-sided [-34.490 to -17.925], Standard Error of Mean 4.168
Statistical Analysis 4: Comparison: Placebo vs Empa 25 mg; Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -27.235, 95% CI 2-sided [-35.586 to -18.884], Standard Error of Mean 4.202

3. Primary Outcome: Change From Baseline in 8-point Glucose
Description: Change from baseline in 8-point glucose to 27 days
Time Frame: baseline and 27 days
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 20 | 19 | 20 | 18 | 17
mg/dL | -17.381 (3.932) | -35.263 (4.121) | -39.867 (3.903) | -43.646 (4.113) | -45.721 (4.187)
Statistical Analysis 1: Comparison: Placebo vs Empa 1 mg; Difference calculated as empa 1mg minus placebo; Test type: Superiority or Other; p = 0.0030, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -17.883, 95% CI 2-sided [-29.529 to -6.236], Standard Error of Mean 5.861
Statistical Analysis 2: Comparison: Placebo vs Empa 5 mg; Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -22.487, 95% CI 2-sided [-33.308 to -11.665], Standard Error of Mean 5.445
Statistical Analysis 3: Comparison: Placebo vs Empa 10 mg; Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -26.265, 95% CI 2-sided [-37.762 to -14.768], Standard Error of Mean 5.785
Statistical Analysis 4: Comparison: Placebo vs Empa 25 mg; Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -28.340, 95% CI 2-sided [-39.665 to -17.015], Standard Error of Mean 5.699

4. Secondary Outcome: Change From Baseline in HbA1c
Description: Change from baseline in HbA1c to 28 days
Time Frame: baseline and 28 days
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 20 | 19 | 20 | 18 | 17
percentage of HbA1c | -0.420 (0.089) | -0.659 (0.093) | -0.717 (0.090) | -0.849 (0.094) | -0.815 (0.096)
Statistical Analysis 1: Comparison: Placebo vs Empa 1 mg; Difference calculated as empa 1mg minus placebo; Test type: Superiority or Other; p = 0.0705, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -0.239, 95% CI 2-sided [-0.498 to -0.020], Standard Error of Mean 0.130
Statistical Analysis 2: Comparison: Placebo vs Empa 5 mg; Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p = 0.0203, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -0.296, 95% CI 2-sided [-0.545 to -0.047], Standard Error of Mean 0.125
Statistical Analysis 3: Comparison: Placebo vs Empa 10 mg; Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p = 0.0014, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -0.429, 95% CI 2-sided [-0.687 to -0.170], Standard Error of Mean 0.130
Statistical Analysis 4: Comparison: Placebo vs Empa 25 mg; Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p = 0.0033, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -0.395, 95% CI 2-sided [-0.654 to -0.135], Standard Error of Mean 0.131

5. Secondary Outcome: Change From Baseline in Fructosamine
Description: Change from baseline in Fructosamine to 28 days
Time Frame: baseline and 28 days
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: umol/L
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 20 | 19 | 20 | 18 | 17
umol/L | -8.436 (12.289) | 4.091 (12.663) | -2.453 (12.362) | -26.294 (12.933) | -28.275 (13.282)
Statistical Analysis 1: Comparison: Placebo vs Empa 1 mg; Difference calculated as empa 1mg minus placebo; Test type: Superiority or Other; p = 0.4823, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = 12.527, 95% CI 2-sided [-22.757 to 47.811], Standard Error of Mean 17.755
Statistical Analysis 2: Comparison: Placebo vs Empa 5 mg; Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p = 0.7305, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = 5.984, 95% CI 2-sided [-28.422 to 40.390], Standard Error of Mean 17.313
Statistical Analysis 3: Comparison: Placebo vs Empa 10 mg; Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p = 0.3213, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -17.858, 95% CI 2-sided [-53.438 to 17.721], Standard Error of Mean 17.903
Statistical Analysis 4: Comparison: Placebo vs Empa 25 mg; Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p = 0.2768, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -19.838, 95% CI 2-sided [-55.869 to 16.192], Standard Error of Mean 18.130

6. Secondary Outcome: Change From Baseline in 1,5-anhydroglucitol
Description: Change from baseline in 1,5-anhydroglucitol to 28 days
Time Frame: baseline and 28 days
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: ug/mL
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 20 | 12 | 11 | 10 | 4
ug/mL | 1.174 (0.439) | -3.018 (0.581) | -3.435 (0.615) | -2.863 (0.622) | -3.713 (0.982)
Statistical Analysis 1: Comparison: Placebo vs Empa 1 mg; Difference calculated as empa 1mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -4.192, 95% CI 2-sided [-5.653 to -2.731], Standard Error of Mean 0.728
Statistical Analysis 2: Comparison: Placebo vs Empa 5 mg; Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -4.609, 95% CI [-6.126 to -3.091], Standard Error of Mean 0.756
Statistical Analysis 3: Comparison: Placebo vs Empa 10 mg; Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -4.036, 95% CI 2-sided [-5.565 to -2.508], Standard Error of Mean 0.762
Statistical Analysis 4: Comparison: Placebo vs Empa 25 mg; Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -4.887, 95% CI 2-sided [-7.048 to -2.726], Standard Error of Mean 1.076

7. Secondary Outcome: Change From Baseline in Fasting Insulin
Description: Change from baseline in Fasting insulin to 28 days
Time Frame: baseline and 28 days
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: uU/mL
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 20 | 19 | 20 | 18 | 17
uU/mL | -0.387 (0.287) | -0.866 (0.295) | -0.766 (0.287) | -1.730 (0.301) | -1.643 (0.312)
Statistical Analysis 1: Comparison: Placebo vs Empa 1 mg; Difference calculated as empa 1mg minus placebo; Test type: Superiority or Other; p = 0.2498, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -0.480, 95% CI 2-sided [-1.302 to 0.343], Standard Error of Mean 0.414
Statistical Analysis 2: Comparison: Placebo vs Empa 5 mg; Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p = 0.3544, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -0.379, 95% CI 2-sided [-1.189 to 0.430], Standard Error of Mean 0.408
Statistical Analysis 3: Comparison: Placebo vs Empa 10 mg; Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p = 0.0018, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -1.343, 95% CI 2-sided [-2.171 to -0.516], Standard Error of Mean 0.416
Statistical Analysis 4: Comparison: Placebo vs Empa 25 mg; Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p = 0.0037, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -1.257, 95% CI 2-sided [-2.094 to -0.419], Standard Error of Mean 0.421

8. Secondary Outcome: Change From Baseline in the Area Under the Curve of Plasma Glucose Levels Until 4 Hours After Intake of a Standardised Food (Meal Tolerance Test)
Description: Change from baseline in the area under the curve of plasma glucose levels until 4 hours after intake of a standardised food (meal tolerance test) to 28 days
Time Frame: baseline and 28 days
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: hr*mg/dL
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 20 | 19 | 20 | 18 | 17
hr*mg/dL | -81.357 (10.481) | -176.771 (10.924) | -190.837 (10.554) | -212.693 (11.023) | -217.698 (11.247)
Statistical Analysis 1: Comparison: Placebo vs Empa 1 mg; Difference calculated as empa 1mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -95.414, 95% CI 2-sided [-125.995 to -64.833], Standard Error of Mean 15.388
Statistical Analysis 2: Comparison: Placebo vs Empa 5 mg; Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -109.480, 95% CI 2-sided [-138.633 to -80.327], Standard Error of Mean 14.670
Statistical Analysis 3: Comparison: Placebo vs Empa 10 mg; Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -131.336, 95% CI 2-sided [-161.848 to -100.824], Standard Error of Mean 15.354
Statistical Analysis 4: Comparison: Placebo vs Empa 25 mg; Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -136.341, 95% CI 2-sided [-166.860 to -105.823], Standard Error of Mean 15.357

9. Secondary Outcome: Change From Baseline in the Area Under the Curve of Glucagon Levels Until 4 Hours After Intake of a Standardised Food (Meal Tolerance Test)
Description: Change from baseline in the area under the curve of glucagon levels until 4 hours after intake of a standardised food (meal tolerance test) to 28 days
Time Frame: baseline and 28 days
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: hr*pg/mL
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 20 | 19 | 20 | 18 | 17
hr*pg/mL | -23.452 (9.177) | -0.785 (9.383) | 7.124 (9.138) | -17.478 (9.635) | -12.437 (9.964)
Statistical Analysis 1: Comparison: Placebo vs Empa 1 mg; Difference calculated as empa 1mg minus placebo; Test type: Superiority or Other; p = 0.0883, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = 22.668, 95% CI 2-sided [-3.470 to 48.805], Standard Error of Mean 13.152
Statistical Analysis 2: Comparison: Placebo vs Empa 5 mg; Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p = 0.0203, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = 30.576, 95% CI 2-sided [4.859 to 56.293], Standard Error of Mean 12.941
Statistical Analysis 3: Comparison: Placebo vs Empa 10 mg; Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p = 0.6541, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = 5.974, 95% CI 2-sided [-20.434 to 32.382], Standard Error of Mean 13.289
Statistical Analysis 4: Comparison: Placebo vs Empa 25 mg; Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p = 0.4206, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = 11.015, 95% CI 2-sided [-16.036 to 38.066], Standard Error of Mean 13.612

10. Secondary Outcome: Change From Baseline in the Area Under the Curve of Insulin Levels Until 4 Hours After Intake of a Standardised Food (Meal Tolerance Test)
Description: Change from baseline in the area under the curve of insulin levels until 4 hours after intake of a standardised food (meal tolerance test) to 28 days
Time Frame: baseline and 28 days
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: hr*uU/mL
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 20 | 19 | 20 | 18 | 17
hr*uU/mL | 2.948 (2.819) | -5.921 (2.896) | -11.396 (2.811) | -12.695 (2.982) | -7.170 (3.048)
Statistical Analysis 1: Comparison: Placebo vs Empa 1 mg; Difference calculated as empa 1mg minus placebo; Test type: Superiority or Other; p = 0.0318, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -8.869, 95% CI 2-sided [-16.949 to -0.789], Standard Error of Mean 4.066
Statistical Analysis 2: Comparison: Placebo vs Empa 5 mg; Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p = 0.0005, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -14.344, 95% CI 2-sided [-22.225 to -6.462], Standard Error of Mean 3.966
Statistical Analysis 3: Comparison: Placebo vs Empa 10 mg; Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -15.642, 95% CI 2-sided [-23.853 to -7.432], Standard Error of Mean 4.131
Statistical Analysis 4: Comparison: Placebo vs Empa 25 mg; Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p = 0.0164, ANCOVA; The baseline value was included as a continuous covariate; Mean Difference (Final Values) = -10.118, 95% CI 2-sided [-18.339 to -1.897], Standard Error of Mean 4.137

11. Secondary Outcome: AUCτ,1
Description: Area under the concentration-time curve of the analyte in plasma after administration of the first dose over a uniform dosing interval τ
Time Frame: Predose and 15 minutes (min), 30min, 45min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 23h55min after first drug administration
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 20 | 19
nmol*h/L | 216 (18.4) | 938 (44.2) | 2040 (19.4) | 5190 (18.6)

12. Secondary Outcome: AUC0-tz
Description: area under the concentration-time curve of the analyte in plasma over the time interval from 0 to last quantifiable plasma concentration
Time Frame: as for outcome 11
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 20 | 19
nmol*h/L | 216 (18.4) | 937 (44.2) | 2040 (19.5) | 5180 (18.6)

13. Secondary Outcome: AUC0-∞
Description: area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 11
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 20 | 19
nmol*h/L | 249 (15.5) | 1070 (44.5) | 2320 (18.1) | 5930 (18.6)

14. Secondary Outcome: Cmax
Description: maximum measured concentration of the analyte in plasma
Time Frame: as for outcome 11
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 20 | 19
nmol/L | 38.5 (28.8) | 166 (47.6) | 358 (29.1) | 844 (15.7)

15. Secondary Outcome: t1/2
Description: terminal half-life of the analyte in plasma
Time Frame: as for outcome 11
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 21 | 20 | 19
hour | 9.55 (14.8) | 9.09 (15.0) | 9.14 (13.3) | 9.26 (15.8)

16. Secondary Outcome: CL/F
Description: apparent clearance of the analyte in plasma after extravascular administration
Time Frame: as for outcome 11
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 20 | 19
mL/min | 149 (15.5) | 173 (44.5) | 159 (18.1) | 156 (18.6)

17. Secondary Outcome: Vz/F
Description: apparent volume of distribution during the terminal phase λz following an extravascular dose
Time Frame: as for outcome 11
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 20 | 19
Liter | 123 (26.1) | 136 (46.3) | 126 (25.5) | 125 (25.3)

18. Secondary Outcome: Ae0-24
Description: amount of the analyte that is eliminated in urine over the time interval 0 to 24
Time Frame: 0-5, 5-12, 12-24 hour after first drug administration
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 18 | 20 | 20 | 19
nmol | 338 (23.7) | 1640 (56.2) | 3460 (17.5) | 8550 (17.0)

19. Secondary Outcome: fe0-24
Description: fraction of the analyte excreted unchanged in urine from time interval 0 to 24
Time Frame: 0-5, 5-12, 12-24 hour after first drug administration
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of Ae0-24 (to dosage)
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 18 | 20 | 20 | 19
percentage of Ae0-24 (to dosage) | 15.2 (23.7) | 14.8 (56.2) | 15.6 (17.5) | 15.4 (17.0)

20. Secondary Outcome: CLR,0-24
Description: renal clearance of the analyte in plasma after extravascular administration - based on 0-24 hours data
Time Frame: Predose and 15 minutes (min), 30min, 45min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 23h55min, 0-5h, 5-12h, 12-24h after first drug administration
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 18 | 19 | 20 | 19
mL/min | 25.7 (21.2) | 28.7 (27.3) | 28.3 (24.4) | 27.5 (23.4)

21. Secondary Outcome: AUCτ,ss
Description: area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ at steady state
Time Frame: Predose and 15 minutes (min), 30min, 45min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h after last drug administration
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 18 | 17
nmol*h/L | 277 (17.0) | 1270 (15.0) | 2580 (17.3) | 6330 (20.3)

22. Secondary Outcome: Cmax,ss
Description: maximum measured concentration of the analyte in plasma at steady state
Time Frame: Predose and 15 minutes (min), 30min, 45min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 36h 48h, 72h after last drug administration
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 18 | 17
nmol/L | 41.4 (32.3) | 182 (31.4) | 393 (28.0) | 836 (29.2)

23. Secondary Outcome: t1/2,ss
Description: terminal half-life of the analyte in plasma at steady state
Time Frame: as for outcome 22
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 18 | 17
hour | 12.2 (45.5) | 11.9 (48.0) | 13.4 (37.7) | 16.4 (48.4)

24. Secondary Outcome: CL/F,ss
Description: apparent clearance of the analyte in plasma after extravascular administration at steady state
Time Frame: as for outcome 22
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 18 | 17
mL/min | 133 (17.0) | 146 (15.0) | 143 (17.3) | 146 (20.3)

25. Secondary Outcome: Vz/F,ss
Description: apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state
Time Frame: as for outcome 22
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 18 | 17
Liter | 141 (37.8) | 151 (48.6) | 166 (43.6) | 208 (51.6)

26. Secondary Outcome: RA,Cmax
Description: accumulation ratios of the analyte in plasma after 28 doses (once daily) over a uniform dosing interval τ, based on Cmax
Time Frame: Predose, 15min, 30min, 45min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 23h55min after first drug administration, and predose, 15min, 30min, 45min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h after last drug administration
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 19 | 18 | 17
ratio | 1.08 (23.3) | 1.07 (54.2) | 1.16 (34.2) | 0.998 (30.4)

27. Secondary Outcome: RA,AUC
Description: accumulation ratios of the analyte in plasma after 28 doses (once daily) over a uniform dosing interval τ, based on AUCτ
Time Frame: as for outcome 26
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 19 | 18 | 17
ratio | 1.28 (9.21) | 1.32 (42.5) | 1.32 (13.1) | 1.23 (12.7)

28. Secondary Outcome: Ae0-24,ss
Description: amount of the analyte that is eliminated in urine at steady state over the time interval 0 to 24
Time Frame: 0-5, 5-12, 12-24 hour after last drug administration
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 18 | 17
nmol | 479 (27.2) | 2250 (44.5) | 4780 (18.6) | 11500 (24.3)

29. Secondary Outcome: fe0-24,ss
Description: fraction of the analyte excreted unchanged in urine at steady state from time interval 0 to 24
Time Frame: 0-5, 5-12, 12-24 hour after last drug administration
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of Ae0-24 (to dosage)
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 18 | 17
percentage of Ae0-24 (to dosage) | 21.6 (27.2) | 20.3 (44.5) | 21.6 (18.6) | 20.8 (24.3)

30. Secondary Outcome: CLR,ss
Description: renal clearance of the analyte at steady state determined over the dosing interval τ
Time Frame: Predose and 15 minutes (min), 30min, 45min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 0-5h, 5-12h, 12-24h after last drug administration
Population: Pharmacokinetic analysis set: all patients who received at least one dose of BI 10773 and had some pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 19 | 20 | 18 | 17
mL/min | 28.8 (25.2) | 29.6 (40.5) | 30.9 (28.1) | 30.3 (28.3)

ADVERSE EVENTS:
Time Frame: Between the first drug administration and the end of the trial after the last drug administration, up to 28 days.
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/19 | 0/21 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 1/21 | 6/19 | 2/21 | 5/20 | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Empa 1 mg (N=19) | Empa 5 mg (N=21) | Empa 10 mg (N=20) | Empa 25 mg (N=19)
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Empa 1 mg (N=19) | Empa 5 mg (N=21) | Empa 10 mg (N=20) | Empa 25 mg (N=19)
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Alpha 1 microglobulin urine increased (Investigations) | 0 | 1 | 0 | 0 | 0
Beta 2 microglobulin urine increased (Investigations) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Additional secondary endpoints were listed in the original protocol. Those endpoints are of exploratory nature only and were not considered relevant for trial conclusions. For more information see tab "Full Text Review", section "More Information".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.